CLINICAL TRIAL: NCT04430699
Title: A Phase 2 Study of Combined Chemo-immunotherapy With Cisplatin-pembrolizumab and Radiation for Unresectable Vulvar Squamous Cell Carcinoma
Brief Title: Cisplatin+Pembrolizumab+RT in Vulvar Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Oladapo O. Yeku,M.D.,Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-109
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Vulvar Cancer; Vulvar Squamous Cell Carcinoma
Keywords: Vulvar Cancer; Vulvar Squamous Cell Carcinoma,; Immunotherapy; Radiation; Pembrolizumab
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Cisplatin; pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab, Cisplatin and Radiation Therapy (Experimental): Treatment period is 36 weeks with 21 day study cycles.
  Participants will receive cisplatin at a predetermined dose 1x weekly, pembrolizumab at a predetermined dose every 3 weeks, concurrently with daily radiation therapy from week 1 up to week 8.
  First 3 participants on the study, may skip 1 or 2 pembrolizumab dosages while receiving radiation therapy.
  Following completion of daily radiation therapy with 1x weekly cisplatin and 1x every 3 weeks pembrolizumab, participants will continue at a pre-determined maintenance dose of pembrolizumab 1x every 3 weeks for a total of 12 cycles or 36 weeks.
  Interventions: Drug: Cisplatin; Drug: Pembrolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — Participants will be given Cisplatin by intravenous infusion at a predetermined dose 1x weekly up to 8 weeks.
  Other Names: Platinol; Platinol-AQ; CDDP
Drug: Pembrolizumab — Participants will be given Pembrolizumab by intravenous infusion at a predetermined dose 1x every 3 weeks up to 36 weeks.
  Other Names: Keytruda
Radiation: Radiation Therapy — Standard of care radiation therapy 1x daily up to 8 weeks.

SUMMARY:
This research is being done to see how well the combination of a standard of care drug, investigational drug, and radiation therapy work against unresectable vulvar squamous cell carcinoma.

This research study involves the following:

* Cisplatin (standard of care drug)
* Pembrolizumab (investigational drug)
* Radiation Therapy (standard of care intervention)

DETAILED DESCRIPTION:
This is a single-arm phase 2 clinical trial involving women with unresectable, incompletely resected, recurrent, or metastatic vulva squamous cell carcinoma. This study combines cisplatin, pembrolizumab, and radiation therapy to see if this combination further increases participants' immune system's efficiency in killing their tumor, and if the combination decreases the chances of participants' cancer coming back.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

This research study involves the following:

* Cisplatin (standard of care drug)
* Pembrolizumab (investigational drug)
* Radiation Therapy (standard of care intervention)

Participants will receive study treatment for up to 36 weeks and will be followed for up to 3 years.

It is expected that about 24 people will take part in this research study.

Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied. The U.S. Food and Drug Administration (FDA) has approved cisplatin as a treatment option for vulva squamous cell carcinoma. The FDA has not approved pembrolizumab for vulva squamous cell carcinoma, but it has been approved for other uses. Cisplatin is a chemotherapy drug and will be given to participants per standard of care.

Radiation therapy will be given to you per standard of care. Pembrolizumab is a drug that may target participants immune systems to increase its efficiency in targeting and killing illnesses and diseases, such as unresectable vulvar squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed unresectable, incompletely resected, recurrent, or metastatic squamous cell carcinoma of the vulva.Patients with unresectable disease are defined as T2 or T3 primary tumors (N0-3, M0) not amenable to surgical resection by standard radical vulvectomy.
* Participants must have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
* Prior therapy: Participants with no prior therapy are eligible and patients with recurrent disease must not have had more than two lines of cytotoxic therapy. Topical or hormonal therapy are not counted towards prior lines. Prior treatment with immunotherapy is allowed, provided treatment was not stopped for grade 2 or greater adverse events.
* Time from prior therapy:

  * Systemic anti-neoplastic therapy: 5 half-lives or 4 weeks, whichever is shorter.
  * Hormonal therapy is not considered anti-neoplastic therapy.
  * Radiotherapy: Any prior irradiation is acceptable provided the site being considered for study has not been previously irradiated.
* Age ≥18 years. Because insufficient dosing or adverse event data are currently available on the use of pembrolizumab in combination with cisplatin-sensitized radiation therapy participants <18 years of age, children are excluded. Vulva cancer is rare in the pediatric population
* ECOG performance status of 0 or 1.
* Participants must have adequate organ and marrow function as defined below (Table 1):

  * Table 1: Adequate Organ Function Laboratory Values

    * Hematological

      * Absolute neutrophil count (ANC) ≥1500/μL
      * Platelets ≥100 000/μL
      * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
    * Renal

      * Creatinine OR Measured or calculated b creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥50 mL/min for participant with creatinine
    * Hepatic

      * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
      * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
    * Coagulation

      * International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
      * ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.
      * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
      * Creatinine clearance (CrCl) should be calculated per institutional standard.
      * Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.
* Participant must be female, and is eligible to participate if she is not pregnant (see Appendix B), not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) as defined in Appendix B OR
  * A WOCBP must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during study treatment, and for at least twelve weeks after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who in the opinion of the investigator cannot safely receive a minimum of 30 Gy in 10 fractions are not eligible for the trial.
* Participants who have received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to first dose of study treatment. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. Re-irradiation to a previously treated site will not be permitted.
* Participants who have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Participants with vulvar melanomas, sarcomas, extramammary Paget's disease, or basal cell carcinoma
* Participants with a history of gastrointestinal or colovesicular fistulae
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Patients with a history of other invasive malignancies, with the exception of nonmelanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required.
* Has a known history of active TB (Bacillus Tuberculosis).
* Pregnant or nursing women are excluded from this study because effects of agents used in this study on infants or the developing human fetus are unknown.
* Presence of other malignancies unless they are considered cured by patient's oncologist.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has a known history of Human Immunodeficiency Virus (HIV).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 36 weeks
  To determine the Overall response rate (ORR) in patients undergoing combination therapy with pembrolizumab and cisplatin-sensitized external beam radiation therapy by RECIST 1.1 criteria.
  This sample size calculation is based on an ORR of greater than or equal to 60%. For recurrent metastatic disease, there are is no standard of care.The ORR estimation is informed by data showing an ORR of 40% in patients with advanced or recurrent metastatic vulvar cancer treated with platinum-based combination therapy. Single agent chemotherapy has an ORR of about 12% (5). Patients with primary disease who are not candidates for upfront surgery have a reported response rates from 55% to 64%.

SECONDARY OUTCOMES:
Recurrence Free Survival (RFS)-6 months | 6 months
  To determine the 6-month Recurrence Free Survival (RFS) in patients with locally advanced, unresectable, or recurrent metastatic vulvar cancer treated with concurrent cisplatin-sensitized radiation therapy and pembrolizumab. A point estimate with exact 95% CI and Kaplan-Meier estimate will be used for the RFS distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Oladapo Yeku, MD, PHD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinical trials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Background] Yeku O, Russo AL, Lee H, Spriggs D. A phase 2 study of combined chemo-immunotherapy with cisplatin-pembrolizumab and radiation for unresectable vulvar squamous cell carcinoma. J Transl Med. 2020 Sep 14;18(1):350. doi: 10.1186/s12967-020-02523-5. PMID 32928237